CLINICAL TRIAL: NCT01012531
Title: Efficacy and Safety of Subcutaneous Cluster Immunotherapy With Cluster-allergoid CLUSTOID Grasses/Rye (Glutaraldehyde-polymerized Allergen Extract of Mixtures of Grass and Rye Allergens) in Patients With Allergic Rhinoconjunctivitis Sensitized to Grass and With or Without Rye Pollen Sensitization
Brief Title: Efficacy and Safety of Specific Immunotherapy With CLUSTOID Grass Pollen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roxall Medizin (Industry)
Responsible Party: Jenny Uhlig, Roxall Medizin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLU-2008-001
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2009-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- highly polymerized allergen extract (Active Comparator)
  Interventions: Biological: Subcutaneous injections with highly polymerized allergen extract
- Placebo (Placebo Comparator)
  Interventions: Biological: Subcutaneous injection with placebo

INTERVENTIONS:
Biological: Subcutaneous injections with highly polymerized allergen extract — cluster schedule
  Arms: highly polymerized allergen extract
Biological: Subcutaneous injection with placebo — cluster schedule
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the efficacy and safety of cluster immunotherapy with highly polymerized allergen extracts.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of allergic rhinitis/rhinoconjunctivitis due to grass and/or rye pollen
* Positive screening skin prick test (wheal diameter > 3 mm)
* Compliance and ability of the patient to complete a Diary Card for self-evaluating of the symptoms and antisymptomatic medication
* Signed and dated patient´s Informed Consent,

Exclusion Criteria:

* Previous immunotherapy with grass and/or rye pollen extracts within the last 3 years,
* Simultaneous participation in other clinical trials,
* Other reasons contra-indicating an inclusion into the trial according to the investigator´s estimation (e.g. poor compliance),
* Auto-immune disorders,
* Severe chronic inflammatory diseases,
* Malignancy,
* Alcohol abuse,
* Existing or intended pregnancy, lactation and/or lack of adequate contraceptive protection,
* Patients being in any relationship or dependency with the sponsor and/or investigator,
* Treatment with beta-blockers (incl. local application) and/or other contra-indicated drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Symptom and medication score | 1 year

SECONDARY OUTCOMES:
Safety of the treatment during the study period | 1 year
Documentation of adverse events | 1 year
Individual symptom scores of the rhinoconjunctivitis symptom score (RSS) during the pollen season | 1 year
Global evaluation and Quality of life questionnaire | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für Rhinologie und Allergologie, Wiesbaden, Germany